CLINICAL TRIAL: NCT07024511
Title: Effectiveness of Auricular Acupuncture for Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Foo Chai Nien, Associate Professor, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024[K]122-01
Record Dates: First submitted 2025-05-23; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Migraine
Keywords: Pain; Migraine
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Acupuncture, Ear; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auricular acupuncture and acupuncture (Experimental): A total of eight treatment sessions will be administered over a period of three weeks, with sessions scheduled approximately every two to three days.
  Interventions: Other: Auricular acupuncture; Other: Acupuncture
- Acupuncture and sham auricular acupuncture (Placebo Comparator): A total of eight treatment sessions will be administered over a period of three weeks, with sessions scheduled approximately every two to three days.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Auricular acupuncture — Auricular acupuncture
  Arms: Auricular acupuncture and acupuncture
Other: Acupuncture — Acupuncture

SUMMARY:
Migraine is a primary headache disorder characterized by recurrent episodes of moderate to severe pain, frequently accompanied by nausea, photophobia, and phonophobia. It ranks as the third most prevalent medical condition globally and is recognized by the World Health Organization (WHO) as one of the top ten causes of disability worldwide. Migraine presents substantial public health concerns due to its considerable socioeconomic burden and its detrimental impact on individuals' quality of life. Although pharmacological treatments are widely available, their effectiveness is often limited, with many patients experiencing inadequate symptom relief or adverse side effects. Consequently, there has been growing interest in non-pharmacological approaches, particularly acupuncture and auricular therapy, due to their favorable safety profiles and reported efficacy in alleviating migraine symptoms. Auricular therapy, a microsystem of acupuncture applied to specific points on the external ear, has gained popularity for its simplicity, low risk, and therapeutic potential. Despite its increasing clinical use, robust scientific evidence supporting the effectiveness of auricular therapy for migraine remains insufficient, underscoring the need for well-designed clinical studies to validate its therapeutic value.

DETAILED DESCRIPTION:
Migraine is a complex and dynamic neurological disorder characterized by fluctuations in attack frequency, duration, severity, and associated symptoms, necessitating timely prevention and effective management strategies. While pharmacological treatments remain the mainstay, their limitations have led to increasing interest in non-pharmacological interventions such as acupuncture. Acupuncture has gained global recognition for its efficacy, particularly in migraine, which is one of the conditions most responsive to this therapy. Supported by strong clinical evidence, acupuncture is considered safe and well-tolerated, with a low incidence of adverse effects. Guidelines for managing primary headache disorders now advocate a range of complementary approaches, including acupuncture, dietary changes, physical activity, and cognitive behavioral therapy which reflecting a paradigm shift towards integrative care. Clinical studies have demonstrated that acupuncture can significantly reduce migraine frequency, shorten attack duration, and alleviate symptom severity. Mechanistic research suggests acupuncture modulates migraine pathophysiology through neuroimmune and neurotransmitter regulation, although further studies are needed to elucidate its molecular effects, particularly beyond the trigeminovascular system. Within Traditional Chinese Medicine, auricular therapy based on stimulating specific points on the external ear aligned with internal organ systems via the "inverted fetus" model offers a simplified, non-invasive modality that activates neural signaling pathways to regulate bodily functions and relieve migraine symptoms. Despite its growing clinical use, further clinical evidence is needed to confirm the therapeutic efficacy and mechanisms of auricular acupuncture in migraine management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having migraine with aura and without aura according to the diagnostic criteria specified by the ICHD 3;
* Aged between 18 and 65 years old;
* Provided written informed consent;
* Headache lasting for 4 to 72 hours and occur at least 5 times (untreated or poorly treated);
* At least 2 out of 4 criteria must be met (unilateral, pulsatile, moderate to severe pain, headache aggravated by daily physical activity, or avoidance of daily activities such as walking or climbing stairs due to headache);
* At least one of the two criteria must be met (nausea and/or vomiting, photophobia, and fear of sound);
* At least one fully recoverable premonitory symptom (visual, sensory, speech and/or language, motor, brainstem, retina); Onset time more than 5 minutes; (8) No prophylaxis treatments with acupuncture or drugs in the past 3 months; (9) Written informed consent provided.

Exclusion Criteria:

* All other diagnoses of chronic, tension-type headache, cluster headache and/or secondary headaches;
* History of psychotic disorder(s).;
* Pregnancy or lactation;
* Severe somatic disorder(s);
* History of severe organic psychiatric disorder(s);
* History of other chronic pain condition(s) in the pass 3 months;
* History of addictive disorder(s);
* Visual Aura Rating Scale, VARS≥5 score;
* Taking long-term painkillers for more than 1 month within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
headache frequency | from baseline to 1 month post treatment.
  The frequency of headaches will be recorded in the form of a headache diary, and doctors will conduct electronic inquiries in WeChat groups every day.

SECONDARY OUTCOMES:
pain severity | from baseline to 1 month post treatment.
  Pain severity is categorized as follows: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). The score is determined by measuring the distance (in millimeters) on a 10 cm line between the "no pain" anchor and the patient's mark using a ruler, providing a score range of 0 to 100.
migraine disability | from baseline to 1 month post treatment
  The Migraine Disability Assessment (MIDAS) questionnaire consists of five questions, each addressing the number of days affected by migraines. The average pain intensity of headaches is rated on a scale from 0 to 10, where 0 indicates no pain and 10 represents the most severe pain.
Change of baseline in the mean quality of life as assessed by Migraine-Specific Quality of Life Questionnaire at 1 month | from baseline to 1 month post treatment
  The Migraine-Specific Quality of Life Questionnaire (MSQ) comprises 3 domains: role function-restrictive (RR), role function-preventive (RP), and emotional function (EF). Each item is scored on a 1-6 scale.
  Raw dimension scores are computed as a sum of item responses and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
physical (physical function, pain intensity)， mental (depression, anxiety, fatigue, sleep disturbance) and social (ability to participate in social roles and activities). | from baseline to 1 month post treatment
  1. Patient-Reported Outcomes Measurement Information System (PROMIS) with 7 PROMIS domains including depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. The total score of each domain is converted to a standardized T score.
  2. In this scale, each item has five response options, with each option scored from 1 to 5 points. For the Anxiety and Depression domains, scoring is reversed: higher scores reflect less severe symptoms. For all other domains, higher scores indicate more severe symptoms or greater impairment. Pain Intensity is rated directly on a 0-10 scale, where 0 represents no pain and 10 represents the worst possible pain.
treatment success | at immediate post treatment
  Patients Global Impression of Improvement (PGI-I) is a transition scale that is a single question asking the patient to rate their condition, as compared with how it is prior to before beginning treatment on a scale. This is measured by success , where it is defined as "very much improved" or "much improved".
red blood cell distribution width (RDW) | from baseline to immediate post treatment
  RDW testing is a part of blood routine and usually does not require special preparation. Patients do not need to be on an empty stomach. To ensure that blood indicators are not affected by time, all patients will have their blood drawn at 10am on the day after the end of treatment
adverse side effects | up to 48 hours after each treatment
  including bleeding, subcutaneous hemorrhage, hematoma, fainting, serious pain, and local infection

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hebei University of Engineering Affiliated Hospital, Handan, Hebei
  - Yurangqiao Community Health Service Center, Xingdong New District, Xingtai City, Xingtai, Hebei

IPD SHARING:
Plan to Share IPD: No